CLINICAL TRIAL: NCT04346108
Title: A Phase 3, Open-label, Non-controlled, Multi-dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability, and Efficacy of Immune Globulin Subcutaneous (Human), 20% Solution (IGSC, 20%) in Japanese Subjects With Primary Immunodeficiency Diseases (PID)
Brief Title: A Study of Immune Globulin Subcutaneous (Human), 20% Solution (IGSC, 20%) in Japanese Participants With Primary Immunodeficiency Diseases (PID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-664-3001; JapicCTI-205162 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Epoch 1: IGIV 200-600 mg/kg (Experimental): Participants received 200 to 600 mg/kg of Immunoglobulin Intravenous (IGIV) infusion for every 3 or 4 weeks for up to 13 weeks.
  Interventions: Biological: Immune Globulin Intravenous (IGIV)
- Epoch 2: IGSC (20%) 50-200 mg/kg (Experimental): Participants who entered to Epoch 2 from Epoch 1 received 50-200 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion once a week up to approximately 24 weeks after Epoch 1.
  Interventions: Biological: Immune Globulin Subcutaneous, 20% Solution (IGSC, 20%)
- Epoch 3: IGSC (20%) 100-400 mg/kg (Experimental): Participants who entered to Epoch 3 from Epoch 1 received 100-400 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion biweekly up to approximately 12 weeks after Epoch 2.
  Interventions: Biological: Immune Globulin Subcutaneous, 20% Solution (IGSC, 20%)

INTERVENTIONS:
Biological: Immune Globulin Intravenous (IGIV) — Participants will receive IGIV infusion.
  Other Names: Immune Globulin Infusion (Human)
  Arms: Epoch 1: IGIV 200-600 mg/kg
Biological: Immune Globulin Subcutaneous, 20% Solution (IGSC, 20%) — Participants will receive IGSC, 20% SC infusion.
  Other Names: Immune Globulin Infusion (Human)
  Arms: Epoch 2: IGSC (20%) 50-200 mg/kg; Epoch 3: IGSC (20%) 100-400 mg/kg

SUMMARY:
In this study, Japanese participants with primary immunodeficiency diseases were treated with Immune Globulin Subcutaneous (Human), 20% solution, (IGSC, 20%). This study will be in 3 parts:

Part 1: Infusions with Immunoglobulin Intravenous (IGIV) every 3 or 4 weeks for 13 weeks.

Part 2: Participants will switch to weekly subcutaneous infusions with IGSC, 20% for 24 weeks.

Part 3: A subset will receive biweekly subcutaneous infusions with IGSC, 20% for 12 weeks.

The main aim of the study is to assess base levels of Immunoglobulin globulin G (IgG) levels in the blood of the participants after weekly and biweekly treatment with IGSC, 20% (in Parts 2 and 3 of the study). Their PID will be treated by their doctor according to their doctor's usual clinical practice.

DETAILED DESCRIPTION:
This study consists of 3 treatment parts (Epoch 1, 2, 3). The total evaluation period of the study will be 57 weeks in which screening period is for 2-8 weeks and Epoch 1 is from Week 8 to Week 21, Epoch 2 is from Week 21 to Week 45, Epoch 3 is from Week 45 to Week 57.

Each participant will receive IGIV treatment in Epoch 1 for a total of 13 weeks, then switch to weekly subcutaneous (SC) treatment with IGSC, 20% in Epoch 2 for a total of 24 weeks and will continue into Epoch 3 for a total of 12 weeks of biweekly SC treatment with IGSC, 20%. Drug dose in Epoch 2 and Epoch 3 will be adjusted so that it will be an equivalent weekly dose of the dose administered in Epoch 1 and twice the dose administrated in Epoch 2 respectively. Epoch 2 will contain two periods, period 1: dose adjustment period (first 12 weeks) and period 2: evaluation period (second 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Be of Japanese descent, defined as born in Japan and having Japanese parents and Japanese maternal and paternal grandparents.
* Participants must have a documented diagnosis of a form of primary humoral immunodeficiency involving antibody formation and requiring gammaglobulin replacement. The diagnosis must be confirmed by the medical director prior to treatment with IGIV.
* Participant is 2 years or older at the time of screening.
* Written informed consent is obtained from either the participants or the participants legally authorized representative prior to any study-related procedures and study product administration.
* Participant has been receiving a consistent dose of IGIV over a period of at least 3 months prior to screening equivalent to approximately 200-600 mg/kg-body weight (BW) per 3- 4 week period, as according to the product package insert
* Participant has a serum trough level of IgG >= 5 gram per liter (g/L) at screening.
* Participant has not had a serious bacterial infection within the 3 months prior to screening.
* Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Participant has a known history of or is positive at screening for one or more of the following: hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for hepatitis C virus (HCV), PCR for human immunodeficiency virus (HIV) Type 1/2.
* Abnormal laboratory values at screening meeting any one of the following criteria (abnormal tests may be repeated once to determine if they are persistent):

  * Persistent alanine aminotransferase (ALT) and aspartate amino transferase (AST) > 2.5 times the upper limit of normal (ULN) for the testing laboratory
  * Persistent severe neutropenia (defined as an absolute neutrophil count [ANC] <= 500/milli cubic meter [mm^3]).
* Participant has presence of renal function impairment defined by estimated glomerular filtration rate (eGFR) is <60 milliliter per minute/ 1.73 square meter (mL/min/1.73m^2).
* Participant has been diagnosed with or has a malignancy (other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix), unless the disease-free period prior to screening exceeds 5 years.
* Participant is receiving anti-coagulation therapy or has a history of thrombotic episodes (including deep vein thrombosis, myocardial infarction, cerebrovascular accident, pulmonary embolism) within 12 months prior to screening or a history of thrombophilia.
* Participant has abnormal protein loss (protein losing enteropathy, nephrotic syndrome).
* Participant has anemia that would preclude phlebotomy for laboratory studies according to standard practice at the site.
* Participant has an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IV immunoglobulin, SC immunoglobulin, and/or Immune Serum Globulin (ISG) infusions.
* Participant has immunoglobulin A (IgA) deficiency (IgA less than 0.07 g/L), known anti IgA antibodies, and a history of hypersensitivity.
* Participant is on preventative (prophylactic) systemic antibacterial antibiotics at doses sufficient to treat or prevent bacterial infections, and cannot stop these antibiotics at the time of screening.
* Participant has active infection and is receiving antibiotic therapy for the treatment of infection at the time of screening.
* Participant has a bleeding disorder, or a platelet count less than 20,000/ microliter (mcL), or, in the opinion of the investigator, would be at significant risk of increased bleeding or bruising as a result of subcutaneous therapy.
* Participant has total protein > 9 gram per deciliter (g/dL) or myeloma, or macroglobulinemia (IgM) or paraproteinemia.
* Women of childbearing potential meeting any one of the following criteria:

  * Participant presents with a positive pregnancy test.
  * Participant is breast feeding.
  * Participant intends to begin nursing during the course of the study.
  * Participant does not agree to employ adequate birth-control measures (e.g. intrauterine device, diaphragm or condom [for male partner] with spermicidal jelly or foam, or birth control pills/patches) throughout the course of the study.
* Participant has participated in another clinical study and has been exposed to an IP or device within 30 days prior to study enrollment.
* Participant is scheduled to participate in another non-observational (interventional) clinical study involving an IP or device during the course of the study.
* Participant has severe dermatitis that would preclude adequate sites for safe product administration.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (8):
- Japan (8):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National Defense Medical College Hospital, Tokorozawa-shi, Saitama
  - Tokyo Medical Dental University Hospital, Bunkyo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in Japan from 11 August 2020 to 22 December 2021.
Pre-assignment Details: Participants diagnosed with primary immunodeficiency diseases (PID) received immunoglobulin administered intravenously (IGIV) in Epoch 1, followed by immunoglobulin administered subcutaneously (IGSC) 20% in Epoch 2 and then followed by Epoch 3 respectively for up to approximately 50 weeks.
Groups:
- Epoch 3: IGSC (20%) 100-400 mg/kg: Participants who entered to Epoch 3 from Epoch 2 received 100-400 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion biweekly up to approximately 12 weeks after Epoch 2.
Period: Epoch 1 (13 Weeks)
Arm/Group | Epoch 1: IGIV 200-600 mg/kg | Epoch 2: IGSC (20%) 50-200 mg/kg | Epoch 3: IGSC (20%) 100-400 mg/kg
Started | 17 | 0 | 0
Completed | 17 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Epoch 2 (24 Weeks After Epoch 1)
Arm/Group | Epoch 1: IGIV 200-600 mg/kg | Epoch 2: IGSC (20%) 50-200 mg/kg | Epoch 3: IGSC (20%) 100-400 mg/kg
Started | 0 | 17 (Those participants who received at least 1 dose of study drug (IGIV) in Epoch 1 and entered Epoch 2.) | 0
Completed | 0 | 15 | 0
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Epoch 3 (12 Weeks After Epoch 2)
Arm/Group | Epoch 1: IGIV 200-600 mg/kg | Epoch 2: IGSC (20%) 50-200 mg/kg | Epoch 3: IGSC (20%) 100-400 mg/kg
Started | 0 | 0 | 7 (Those participants who received at least 1 dose of study drug (IGIV or IGSC) in Epoch 1 and Epoch 2 entered Epoch 3.)
Completed | 0 | 0 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Groups:
- IGIV 200 to 600 mg/kg + IGSC [50 to 200 and 100 to 400] mg/kg: Participants received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks up to 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
Arm/Group | IGIV 200 to 600 mg/kg + IGSC [50 to 200 and 100 to 400] mg/kg
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (21.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 48.16 (18.120)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 152.15 (20.076)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated as [weight (kg) / height(m)^2]
  kg/m^2 | 19.88 (3.242)

OUTCOME MEASURES:

1. Primary Outcome: Epoch 2: Total Serum Trough Levels of Immune Globulin G (IgG) Antibodies During Period 2
Description: Total serum trough levels of IgG antibodies measured during period 2 of Epoch 2 were assessed.
Time Frame: Epoch 2 (period 2): Up to 24 weeks
Population: Pharmacokinetic Analysis Set (PKAS) 1 included all participants in the all-treated set who have had at least 1 evaluable serum IgG concentration value and have had no major protocol deviations or events that would affect the serum IgG concentration analysis results. Only PKAS 1 participants in Epoch 2 were analyzed for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: grams per liter (g/L)
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 17
grams per liter (g/L) | 8.56 [8.03 to 9.12]

2. Primary Outcome: Epoch 3: Total Serum Trough Levels of IgG Antibodies
Description: Total serum trough levels of IgG antibodies measured during Epoch 3 were assessed.
Time Frame: Epoch 3: Up to Week 12
Population: PKAS 1 included all participants in the all-treated set who have had at least 1 evaluable serum IgG concentration value and have had no major protocol deviations or events that would affect the serum IgG concentration analysis results. Only PKAS 1 participants in Epoch 3 were analyzed for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | Epoch 3: IGSC (20%) 100-400 mg/kg
Number analyzed (Participants) | 7
g/L | 8.39 [7.89 to 8.91]

3. Secondary Outcome: Epoch 1: Total Serum Trough Levels of IgG Antibodies
Description: Total serum trough levels of IgG antibodies measured during Epoch 1 were assessed.
Time Frame: Epoch 1: Up to Week 13
Population: PKAS 1 included all participants in the all-treated set who have had at least 1 evaluable serum IgG concentration value and have had no major protocol deviations or events that would affect the serum IgG concentration analysis results. Only PKAS 1 participants in Epoch 1 were analyzed for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Groups:
- Epoch 1: IGIV 200-600 mg/kg: Participants received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for up to 13 weeks.
Arm/Group | Epoch 1: IGIV 200-600 mg/kg
Number analyzed (Participants) | 17
g/L | 8.18 [7.71 to 8.68]

4. Secondary Outcome: Epoch 2: Area Under the Curve From Time 0 to Last Interval (AUC0-last) for Total Serum Levels of IgG
Time Frame: Epoch 2: Week 21
Population: PKAS 2 included all participants >=12 years of age in the all-treated set who have had at least 1 evaluable serum IgG concentration value during Epoch 2 and have had no major protocol deviations or events that would affect the serum IgG concentration analysis results. Overall number analyzed are the number of participants with data available for analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: g*day/L
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
g*day/L | 58.9 [48.7 to 71.3]

5. Secondary Outcome: Epoch 2: AUC0-last for Total Serum Levels of IgG Subclasses
Description: Total serum levels of IgG subclasses IgG 1, IgG 2, IgG 3, and IgG 4 were determined.
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: g*day/L
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
g*day/L
  IgG 1 | 35.8 [32.4 to 39.5]
  IgG 2 | 23.4 [20.4 to 26.9]
  IgG 3 | 1.32 [0.624 to 2.80]
  IgG 4 | 1.67 [1.10 to 2.53]

6. Secondary Outcome: Epoch 2: Apparent Clearance (CL/F) for Total Serum Levels of IgG
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg/day
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
mL/kg/day | 1.93 [1.71 to 2.19]

7. Secondary Outcome: Epoch 2: CL/F for Total Serum Levels of IgG Subclasses
Description: Total serum levels of IgG subclasses IgG 1, IgG 2, IgG 3, and IgG 4 were determined.
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg/day
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
mL/kg/day
  IgG 1 | 3.18 [2.88 to 3.51]
  IgG 2 | 4.86 [4.18 to 5.66]
  IgG 3 | 99.5 [37.1 to 266]
  IgG 4 | 68.3 [48.3 to 96.6]

8. Secondary Outcome: Epoch 2: Maximum Concentration (Cmax) for Total Serum Levels of IgG
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
g/L | 9.08 [7.46 to 11.1]

9. Secondary Outcome: Epoch 2: Cmax for Total Serum Levels of IgG Subclasses
Description: Total serum levels of IgG subclasses IgG 1, IgG 2, IgG 3, and IgG 4 were determined.
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
g/L
  IgG 1 | 5.40 [4.95 to 5.89]
  IgG 2 | 3.51 [3.06 to 4.03]
  IgG 3 | 0.202 [0.0960 to 0.425]
  IgG 4 | 0.256 [0.169 to 0.387]

10. Secondary Outcome: Epoch 2: Minimum Concentration (Cmin) for Total Serum Levels of IgG
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
g/L | 7.45 [6.17 to 8.99]

11. Secondary Outcome: Epoch 2: Cmin for Total Serum Levels of IgG Subclasses
Description: Total serum levels of IgG subclasses IgG 1, IgG 2, IgG 3, and IgG 4 were determined.
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
g/L
  IgG 1 | 4.89 [4.34 to 5.51]
  IgG 2 | 3.15 [2.70 to 3.68]
  IgG 3 | 0.181 [0.0861 to 0.381]
  IgG 4 | 0.218 [0.153 to 0.311]

12. Secondary Outcome: Epoch 2: Time to Maximum Concentration (Tmax) for Total Serum Levels of IgG
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
hours | 71.08 [22.82 to 168.23]

13. Secondary Outcome: Epoch 2: Tmax for Total Serum Levels of IgG Subclasses
Description: Total serum levels of IgG subclasses IgG 1, IgG 2, IgG 3, and IgG 4 were determined.
Time Frame: Epoch 2: Week 21
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Epoch 2: IGSC (20%) 50-200 mg/kg
Number analyzed (Participants) | 7
hours
  IgG 1 | 71.08 [22.82 to 118.80]
  IgG 2 | 71.08 [0.00 to 164.32]
  IgG 3 | 72.92 [71.08 to 118.80]
  IgG 4 | 71.17 [70.13 to 118.80]

14. Secondary Outcome: Trough Levels of Specific Antibodies to Clinically Relevant Pathogens: Clostridium Tetani Toxoid and Hepatitis B Virus (HBV)
Description: Trough levels of specific antibodies to clinically relevant pathogen (Clostridium tetani toxoid and HBV) were assessed in Epoch 1, Epoch 2 and Epoch 3. Data was analyzed per interval in each Epoch for this outcome measure.
Time Frame: Epoch 1 (Week 1); Epoch 2 (Week 1, 24); Epoch 3 (Week 1, 13)
Population: PKAS 1 included all participants in the all-treated set who have had at least 1 evaluable serum IgG concentration value and have had no major protocol deviations or events that would affect the serum IgG concentration analysis results. Overall number analyzed are the number of participants available for analyses. Data is represented as per doses received for specific interval in each Epoch for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU)/mL
Groups:
- Epoch 1: IGIV 3-week Interval (Week 1): Participants received 200 to 600 mg/kg of Immunoglobulin Intravenous (IGIV) infusion for every 3 weeks for up to 13 weeks.
- Epoch 1: IGIV 4-week Interval (Week 1): Participants received 200 to 600 mg/kg of Immunoglobulin Intravenous (IGIV) infusion for every 4 weeks for up to 13 weeks.
- Epoch 2: IGSC, 20% Weekly (Week 1): Participants who entered to Epoch 2 from Epoch 1 received 50-200 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion once a week up to approximately 24 weeks after Epoch 1.
- Epoch 2: IGSC, 20% Weekly (EOS [Week 24]/ET): Participants who entered to Epoch 2 from Epoch 1 received 50-200 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion once a week up to end of study (EOS) (24 weeks) or early termination (ET) after Epoch 1.
- Epoch 3: IGSC, 20% Biweekly (Week 1); Epoch 3: IGSC, 20% Biweekly (Week 13): Participants who entered to Epoch 3 from Epoch 2 received 100-400 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion biweekly up to EOS (13 weeks) after Epoch 2.
Arm/Group | Epoch 1: IGIV 3-week Interval (Week 1) | Epoch 1: IGIV 4-week Interval (Week 1) | Epoch 2: IGSC, 20% Weekly (Week 1) | Epoch 2: IGSC, 20% Weekly (EOS [Week 24]/ET) | Epoch 3: IGSC, 20% Biweekly (Week 1) | Epoch 3: IGSC, 20% Biweekly (Week 13)
Number analyzed (Participants) | 5 | 12 | 17 | 10 | 7 | 7
International units (IU)/mL
  Clostridium Tetani Toxoid | 0.524 [0.290 to 0.949] | 0.602 [0.364 to 0.997] | 0.674 [0.468 to 0.970] | 1.52 [1.11 to 2.08] | 1.97 [1.65 to 2.35] | 1.80 [1.35 to 2.39]
  Hepatitis B Virus | 27.7 [17.8 to 43.0] | 35.2 [17.5 to 70.9] | 54.1 [33.7 to 87.0] | 486 [335 to 706] | 645 [452 to 920] | 923 [832 to 1020]

15. Secondary Outcome: Trough Levels of Specific Antibodies to Clinically Relevant Pathogen: Haemophilus Influenzae (HIB)
Description: Trough levels of specific antibodies to clinically relevant pathogens (HIB) were assessed in Epoch 1, Epoch 2, and Epoch 3. Data was analyzed per interval in each Epoch for this outcome measure.
Time Frame: Epoch 1 (Week 1); Epoch 2 (Week 1, 24); Epoch 3 (Week 1, 13)
Population: PKAS 1 included all participants in the all-treated set who have had at least 1 evaluable serum IgG concentration value and have had no major protocol deviations or events that would affect the serum IgG concentration analysis results. Overall number analyzed are the number of participants available for analyses. Data is represented as per doses received for specific intervals in each Epoch for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Groups:
- Epoch 2: IGSC, 20% Weekly (EOS [Week 24]/ET): Participants who entered to Epoch 2 from Epoch 1 received 50-200 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion once a week up to EOS (24 weeks) or ET after Epoch 1.
Arm/Group | Epoch 1: IGIV 3-week Interval (Week 1) | Epoch 1: IGIV 4-week Interval (Week 1) | Epoch 2: IGSC, 20% Weekly (Week 1) | Epoch 2: IGSC, 20% Weekly (EOS [Week 24]/ET) | Epoch 3: IGSC, 20% Biweekly (Week 1) | Epoch 3: IGSC, 20% Biweekly (Week 13)
Number analyzed (Participants) | 5 | 12 | 17 | 10 | 7 | 7
mg/L | 1.58 [0.568 to 4.38] | 1.55 [1.11 to 2.18] | 2.50 [1.95 to 3.20] | 1.77 [1.07 to 2.91] | 2.04 [1.74 to 2.39] | 1.73 [1.46 to 2.04]

16. Secondary Outcome: Health Related Quality of Life: Treatment Preference
Description: Treatment preference questionnaire is a self-administered questionnaire developed to assess participants' preference towards the administration of new IGSC therapy. There are 4-items on the questionnaire, which investigate a participant's preference on the clinic/hospital/home setting of receiving the immunoglobulin therapy, the participant's rating on the frequency and method of administration, and the participant's preference to continue receiving the IGSC treatment. The questionnaire included following categories: Where do you prefer to receive your immunoglobulin therapy, The frequency of administration, as pre-specified in protocol, data is reported as per age (2-13 years and >=14 years).
Time Frame: Up to approximately 1.5 years
Population: All-Treated Set included all enrolled participants of age '2-13 years' and '>=14 years' who received at least 1 dose of study drug (IGIV or IGSC). Number analyzed is the number of participants with data available for analyses at specific timepoints.
Measure: Count of Participants; unit: Participants
Groups:
- IGSC: Epoch 2: 2-13 Years: Participants aged 2-13 years received approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2.
- IGSC: Epoch 2: >=14 Years: Participants aged >=14 years received approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2.
- IGSC: Epoch 3: 2-13 Years: Participants aged 2-13 years received approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
- IGSC: Epoch 3: >=14 Years: Participants aged >=14 years received approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
Arm/Group | IGSC: Epoch 2: 2-13 Years | IGSC: Epoch 2: >=14 Years | IGSC: Epoch 3: 2-13 Years | IGSC: Epoch 3: >=14 Years
Number analyzed (Participants) | 4 | 6 | 2 | 5
Participants
  Where do you Prefer to Receive Your Immunoglobulin Therapy: At Hospital | 0 | 0 | 0 | 1
  Where do you Prefer to Receive Your Immunoglobulin Therapy: At Home | 3 | 1 | 1 | 4
  Where do you Prefer to Receive Your Immunoglobulin Therapy: No Preference | 1 | 5 | 1 | 0
  The Frequency of Administration: Like Very Much | 2 | 1 | 1 | 4
  The Frequency of Administration: Like | 1 | 3 | 1 | 1
  The Frequency of Administration: No Preference | 1 | 2 | 0 | 0
  The Frequency of Administration: Dislike Very Much | 0 | 1 | 0 | 0

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs was defined as adverse events (AEs) with onset after date-time of first dose of study drug, or medical conditions present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. Any TEAE that is recorded by the investigator as "possibly related" or "probably related" to IP was considered as IGSC, 20%-related AE, and any AE recorded as "unlikely related" or "not related" was considered as unrelated AE. AEs included vital signs, clinical laboratory measurements.
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Count of Participants; unit: Participants
Groups:
- Epoch 1: Immune Globulin Intravenous (IGIV): Participants received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for up to 13 weeks.
- Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC): Participants who entered to Epoch 2 from Epoch 1 received 50-200 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion once a week up to approximately 24 weeks after Epoch 1.
- Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC): Participants who entered to Epoch 3 from Epoch 2 received 100-400 mg/kg of Immune Globulin Subcutaneous (Human) 20% infusion biweekly up to approximately 12 weeks after Epoch 2.
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
Participants | 11 | 16 | 3

18. Secondary Outcome: Number of Participants With Tolerability Events Related to the Infusion of Study Drug
Description: An infusion is considered tolerable if the infusion rate was not reduced, or the infusion was not interrupted or stopped, due to TEAE related to study drug (IGIV or IGSC) infusion. A tolerability event is considered to have occurred if an infusion was not tolerable in Epoch 1, Epoch 2 and Epoch 3. Number of participants with tolerability events related to infusion of IP were assessed.
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
Participants
  Infusions With Infusion Rate Reduced | 0 | 0 | 0
  Infusions That Were Interrupted | 0 | 1 | 0
  Infusions That Were Stopped | 0 | 0 | 0
  Infusions With Infusion Rate Reduced or Interrupted or Stopped | 0 | 1 | 0

19. Secondary Outcome: Annual Rate of Validated Acute Serious Bacterial Infections (ASBI)
Description: The ASBI rate was calculated as the mean number of acute serious bacterial infections per participants per year. Annual rate of validated acute serious bacterial infections per participant was assessed.
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Mean (Standard Deviation); unit: number of infections per year
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
number of infections per year | 0.0 (0.00) | 0.25 (1.042) | 0.0 (0.00)

20. Secondary Outcome: Annual Rate of All Infections Per Year
Description: Annual rate is the number of participants reporting any infection per year.
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Mean (Standard Deviation); unit: number of infections per year
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
number of infections per year | 1.65 (2.479) | 2.78 (3.074) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 1.65, 95% CI 2-sided [0.73 to 3.15]
Statistical Analysis 2: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 0.00, 95% CI 2-sided [0.00 to 0.00]
Statistical Analysis 3: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 2.48, 95% CI 2-sided [1.34 to 4.13]

21. Secondary Outcome: Number of Days Participants Not Able to Attend School or Work to Perform Normal Daily Activities Due to Illness/Infection
Description: Number of days not able to attend school or work to perform normal daily activities due to illness/infection are standardized per year (365.25 days). The number of days not able to attend school or work to perform normal daily activities due to illness/infection were assessed.
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Median (Full Range); unit: days
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
days | 0.00 [0.0 to 16.1] | 0.00 [0.0 to 17.2] | 4.30 [0.0 to 38.7]
Statistical Analysis 1: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 2.60, 95% CI 2-sided [1.02 to 5.30]
Statistical Analysis 2: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 9.82, 95% CI 2-sided [2.82 to 23.82]
Statistical Analysis 3: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 2.87, 95% CI 2-sided [1.37 to 5.18]

22. Secondary Outcome: Number of Days Participants Were on Antibiotics
Description: Number of days on antibiotics is defined as the number of days those antibiotics were taken as concomitant medications and is standardized to per year (365.25 days). Antibiotics are defined as any medication under anatomical therapeutic chemical Level 2 therapeutic class "ANTIBACTERIALS FOR SYSTEMIC USE". If a participant took multiple antibiotics on a single day, that day is counted for only once. Protocol defined prophylactic antibiotics for viral, fungal or protozoal infections (e.g. trimethoprim/sulfamethoxazole twice a week for pneumocystis) which are not treated by immunoglobulin, were excluded from this analysis.
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Median (Full Range); unit: days
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
days | 0.00 [0.0 to 31.8] | 0.00 [0.0 to 34.5] | 0.00 [0.0 to 21.5]
Statistical Analysis 1: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 4.01, 95% CI [1.46 to 8.54]
Statistical Analysis 2: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 3.07, 95% CI 2-sided [0.37 to 10.74]
Statistical Analysis 3: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 5.87, 95% CI 2-sided [2.32 to 11.93]

23. Secondary Outcome: Number of Participants Hospitalized Due to Illness or Infection
Description: Number of participants with hospitalization are standardized to per year (365.25 days). A hospitalization is counted for a specific epoch only if that hospitalization started during that epoch.
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
Participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 0.00, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 2: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 0.13, 95% CI 2-sided [0.03 to 0.35]
Statistical Analysis 3: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 0.00, 95% CI 2-sided [0.00 to 0.00]

24. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay per stay is standardized to per year (365.25 days). A hospitalization is counted for a specific epoch only if that hospitalization started during that epoch.
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Median (Full Range); unit: days
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
days | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 17.4] | 0.00 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 0.00, 95% CI 2-sided [0.00 to 0.00]
Statistical Analysis 2: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 1.04, 95% CI 2-sided [0.25 to 2.76]

25. Secondary Outcome: Number of Acute Physician Visits Due to Illness/Infection
Description: Number of acute physician visits is standardized to per year (365.25 days).
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Population: All-Treated Set included all enrolled participants who received at least 1 dose of study drug (IGIV or IGSC).
Measure: Mean (Standard Deviation); unit: number of visits per year
Arm/Group | Epoch 1: Immune Globulin Intravenous (IGIV) | Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) | Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC)
Number analyzed (Participants) | 17 | 17 | 7
number of visits per year | 1.18 (3.098) | 3.30 (6.807) | 1.624 (8.121)
Statistical Analysis 1: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 1.18, 95% CI 2-sided [0.38 to 2.68]
Statistical Analysis 2: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 2.35, 95% CI 2-sided [0.91 to 4.82]
Statistical Analysis 3: Comparison: Epoch 1: Immune Globulin Intravenous (IGIV) vs Epoch 2: Immune Globulin Subcutaneous 20% Solution (IGSC) vs Epoch 3: Immune Globulin Subcutaneous 20% Solution (IGSC); Test type: Superiority; Poisson Estimate = 0.61, 95% CI 2-sided [0.07 to 2.15]

26. Secondary Outcome: Health-related Quality of Life (HRQoL): Pediatric Quality of Life Inventory (PedsQL) Total Scale Score
Description: Peds-QL=generic HR QoL instrument designed specifically for pediatrics has domains as:general health/activities,feelings/emotional,social functioning,school functioning.In this study,2-7 years (parent as observer),8-13 years (participant as observer) for Peds-QL health questionnaire was analyzed.Higher scores=better QOL for all domains.This modular instrument used 5-point scale:0(never) to 4(almost always).Items are reversed scored;linearly transformed to 0-100 scale as follows:0=100,1=75,2=50,3=25,4=0.4 dimensions(physical, emotional, social, & school functioning) are scored.PEDS-QL Total Scale Score has 0-100 scale,higher scores=better HRQoL.
Time Frame: Baseline up to end of study (approximately 1.5 years)
Population: All-Treated Set included all enrolled participants of age group '2-7 years' and '8-13 years' who received at least 1 dose of study drug (IGIV or IGSC). Number analyzed are the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Age 2-7 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]: Participants aged 2-7 years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
- Age 8-13 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]: Participants aged 8-13 years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
Arm/Group | Age 2-7 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg] | Age 8-13 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]
Number analyzed (Participants) | 2 | 4
score on a scale
  IGIV: Epoch 1: Baseline (Week 1) | 88.04 (13.835) | 87.23 (11.820)
  IGSC: Epoch 2: Change from Baseline (Week 1) | 9.78 (15.372) | -6.79 (9.977)
  IGSC: Epoch 3: Change from Baseline (Week 1): number analyzed (Participants) | 1 | 1
  IGSC: Epoch 3: Change from Baseline (Week 1) | 14.13 (NA) — Standard deviation was not estimable for 1 participant | 20.65 (NA) — Standard deviation was not estimable due to 1 participant.
  IGSC: Epoch 3: Change from Baseline (EOS/ET]) | 3.26 (7.686) | 4.08 (16.374)

27. Secondary Outcome: EuroQoL (Quality of Life)-5 Dimensions 3 Levels (EQ-5D-3L) Total Scale Score
Description: EQ-5D-3L health questionnaire=participant answered questionnaire scoring 5 dimensions -mobility,self-care,usual activities, pain/discomfort and anxiety/depression. n this study, 2-11 years (parent as observer),12 years and older (participant as observer) for EQ-5D-3L health questionnaire was analyzed.Health state index score range from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome.EQ visual analogue scale range from 0 to 100, where higher scores indicate better health status.Data is reported as per age groups (2-11 years and >=12 years).
Time Frame: Baseline up to end of the study (approximately 1.5 years)
Population: All-Treated Set included all enrolled participants of age group '2-11 years' and '>=12 years' who received at least 1 dose of study drug (IGIV or IGSC). Number analyzed is the number of participants with data available for analyses at specific timepoints
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Age 2-11 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]: Participants aged 2-11 years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
- Age >=12 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]: Participants aged >=12 years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
Arm/Group | Age 2-11 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg] | Age >=12 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]
Number analyzed (Participants) | 4 | 13
score on a scale
  IGIV: Epoch 1: Baseline (Week 1): Health State Index Score | 0.8080 (0.04619) | 0.8217 (0.04544)
  IGIV: Epoch 1: Baseline (Week 1): EQ Visual Analogue Scale | 87.5 (15.55) | 77.1 (22.16)
  IGSC: Epoch 2: Change from Baseline (Week 1): Health State Index Score: number analyzed (Participants) | 3 | 13
  IGSC: Epoch 2: Change from Baseline (Week 1): Health State Index Score | -0.0270 (0.12275) | 0.0016 (0.03318)
  IGSC: Epoch 2: Change from Baseline (Week 1): EQ Visual Analogue Scale: number analyzed (Participants) | 3 | 13
  IGSC: Epoch 2: Change from Baseline (Week 1): EQ Visual Analogue Scale | -5.0 (5.00) | 4.2 (17.15)
  IGSC: Epoch 3: Change from Baseline (Week 1): Health State Index Score: number analyzed (Participants) | 1 | 6
  IGSC: Epoch 3: Change from Baseline (Week 1): Health State Index Score | 0.0000 (NA) — Standard deviation was not estimable for 1 participant | 0.0133 (0.03266)
  IGSC:Epoch 3: Change from Baseline (Week 1): EQ Visual Analogue Scale: number analyzed (Participants) | 1 | 6
  IGSC:Epoch 3: Change from Baseline (Week 1): EQ Visual Analogue Scale | 0.0 (NA) — Standard deviation was not estimable for 1 participant | -1.3 (12.39)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Health State Index Score | 0.0400 (0.04619) | 0.0229 (0.04566)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): EQ Visual Analogue Scale | 1.3 (6.29) | 6.9 (13.21)

28. Secondary Outcome: Health-related Quality of Life (HRQoL): Short Form-36 Health Survey (SF-36) Score
Description: SF-36=generic quality-of-life instrument that has been widely used to assess HRQL of participants.In this study, 14 years and older (participant as observer) for SF-36 health questionnaire was analyzed. Generic instruments are used in general populations to assess a wide range of domains applicable to a variety of health states, conditions, and diseases.SF-36=36 items aggregated into 8 multi-item scales (physical functioning, role - physical, bodily pain, general health, vitality, social functioning, role - emotional, and mental health), with scores ranging from 0 to 100.Higher scores=better HRQL. As pre-specified in protocol data is reported for participants with age group of 14 years or older.
Time Frame: Baseline up to end of the study (approximately 1.5 years)
Population: All-Treated Set included all enrolled participants of age '14 years and above' who received at least 1 dose of study drug (IGIV or IGSC). Number analyzed is the number of participants with data available for analyses at specific timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Age 14 Years and Above: IGIV 200 to 600 mg/kg + IGSC (20%) 50 to 200 mg/kg and 100 to 400 mg/kg: Participants aged 14 and above years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
Arm/Group | Age 14 Years and Above: IGIV 200 to 600 mg/kg + IGSC (20%) 50 to 200 mg/kg and 100 to 400 mg/kg
Number analyzed (Participants) | 11
score on a scale
  IGIV: Epoch 1: Baseline (Week 1): Physical Component Summary Score | 50.21 (7.282)
  IGIV: Epoch 1: Baseline (Week 1): Mental Component Summary Score | 50.59 (8.114)
  IGSC: Epoch 2: Change from Baseline (Week 1): Physical Component Summary Score | 0.10 (7.142)
  IGSC: Epoch 2: Change from Baseline (Week 1): Mental Component Summary Score | -0.30 (2.294)
  IGSC: Epoch 3: Change from Baseline (Week 1): Physical Component Summary Score: number analyzed (Participants) | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Physical Component Summary Score | 1.81 (8.189)
  IGSC: Epoch 3: Change from Baseline (Week 1): Mental Component Summary Score: number analyzed (Participants) | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Mental Component Summary Score | 3.60 (5.352)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Physical Component Summary Score: number analyzed (Participants) | 10
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Physical Component Summary Score | 0.23 (4.649)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Mental Component Summary Score: number analyzed (Participants) | 10
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Mental Component Summary Score | 4.32 (8.185)

29. Secondary Outcome: Health Related Quality of Life: Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) Score
Description: TSQM=is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. In this study, 2-12 years (parent as observer), 13 years and older (participant as observer) for TSQM health questionnaire will be analyzed. TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are effectiveness, convenience, and global satisfaction. The score of each of the 3 domains is based on an algorithm to create a score of 0 to 100. Higher score indicated greater satisfaction in that domain. As pre-specified in protocol, data is reported as per age group (2-12 years and >=13 years).
Time Frame: Baseline up to end of the study (approximately 1.5 years)
Population: All-Treated Set included all enrolled participants of age group ' 2-12 years' and '>=3 years' who received at least 1 dose of study drug (IGIV or IGSC). Number analyzed is the number of participants with data available for analyses at specific timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Age 2-12 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]: Participants aged 2-12 years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
- Age >=13 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]: Participants aged >=13 years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
Arm/Group | Age 2-12 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg] | Age >=13 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]
Number analyzed (Participants) | 6 | 11
score on a scale
  IGIV: Epoch 1: Baseline (Week 1): Effectiveness | 69.44 (14.380) | 75.25 (18.817)
  IGIV: Epoch 1: Baseline (Week 1): Convenience | 62.96 (13.907) | 65.66 (23.016)
  IGIV: Epoch 1: Baseline (Week 1): Global Satisfaction | 75.00 (17.928) | 74.68 (18.173)
  IGSC: Epoch 2: Change from Baseline (Week 1): Effectiveness: number analyzed (Participants) | 5 | 11
  IGSC: Epoch 2: Change from Baseline (Week 1): Effectiveness | 2.22 (9.296) | -1.52 (10.568)
  IGSC: Epoch 2: Change from Baseline (Week 1): Convenience: number analyzed (Participants) | 5 | 11
  IGSC: Epoch 2: Change from Baseline (Week 1): Convenience | 3.33 (16.942) | 5.05 (13.484)
  IGSC: Epoch 2: Change from Baseline (Week 1): Global Satisfaction: number analyzed (Participants) | 5 | 11
  IGSC: Epoch 2: Change from Baseline (Week 1): Global Satisfaction | -2.86 (10.833) | 1.30 (10.507)
  IGSC: Epoch 3: Change from Baseline (Week 1): Effectiveness: number analyzed (Participants) | 2 | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Effectiveness | 2.78 (3.928) | -10.00 (52.673)
  IGSC: Epoch 3: Change from Baseline (Week 1): Convenience: number analyzed (Participants) | 2 | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Convenience | 13.89 (19.642) | 15.56 (12.669)
  IGSC: Epoch 3: Change from Baseline (Week 1): Global Satisfaction: number analyzed (Participants) | 2 | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Global Satisfaction | -7.14 (10.02) | 4.29 (29.709)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Effectiveness | 9.26 (10.924) | 6.57 (18.892)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Convenience | 5.56 (22.222) | 9.09 (23.210)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Global Satisfaction | 7.14 (23.905) | 3.90 (23.768)

30. Secondary Outcome: Health Related Quality of Life: Treatment Satisfaction Questionnaire for Life Quality Index (LQI) Score
Description: LQI=self-administered questionnaire developed specifically for participants/legal guardians involved in IGIV treatments.2-13 years (parent as observer),14 years and older (participant as observer) for LQI health questionnaire was analyzed.LQI=15-items, divided into 4 domains: treatment interferences(TI)[6 items],therapy-related problems(TRP)[4 items],therapy setting(TS)[3 items];treatment costs(TC)[2 items].Items are rated on a 7-point Likert-type scale ranging from 1:"Extremely bad" to 7:"Extremely good".Total scores=0 to 100,higher scores=highest possible satisfaction with factors such as independence,therapy convenience,social/school/work activities;health and travel costs.As pre-specified in protocol, data is reported as per age (2-13 years and >=14 years).All-Treated Set included all enrolled participants of age group '2-13 years' and '>=14 years' who received at least 1 dose of study drug (IGIV or IGSC).'n'=Number analysed are participants with data available for analysis.
Time Frame: Baseline up to end of the study (approximately 1.5 years)
Population: All-Treated Set included all enrolled participants of age group '2-13 years' and '>=14 years' who received at least 1 dose of study drug (IGIV or IGSC). Number analyzed is the number of participants with data available for analyses at specific timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Age 2-13 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]: Participants aged 2-13 years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
- Age >=14 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]: Participants aged >=14 years received 200 to 600 mg/kg of IGIV infusion for every 3 or 4 weeks for a total of 13 weeks in Epoch 1; followed by approximately 50 to 200 mg/kg of IGSC infusion,20% once a week for a total of 24 weeks after Epoch 1 in Epoch 2; followed by approximately 100 to 400 mg/kg of IGSC infusion, 20% once every two weeks for a total of 12 weeks after Epoch 2 in Epoch 3.
Arm/Group | Age 2-13 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg] | Age >=14 Years: Epoch 1[IGIV 200-600 mg/kg]+Epoch 2 [IGSC 50-100 mg/kg]+Epoch 3 [IGSC 100-400 mg/kg]
Number analyzed (Participants) | 6 | 11
score on a scale
  IGIV: Epoch 1: Baseline (Week 1): Factor 1 Treatment Interference | 81.48 (14.873) | 77.02 (17.963)
  IGIV: Epoch 1: Baseline (Week 1): Factor 2 Therapy-Related Problems | 81.94 (15.516) | 79.17 (15.811)
  IGIV: Epoch 1: Baseline (Week 1): Factor 3 Therapy Setting | 77.78 (20.488) | 74.75 (23.748)
  IGIV: Epoch 1: Baseline (Week 1): Factor 4 Treatment Costs | 65.28 (24.391) | 53.79 (21.847)
  IGSC: Epoch 2: Change from Baseline (Week 1): Factor 1 Treatment Interference | -8.33 (21.445) | -2.53 (14.351)
  IGSC: Epoch 2: Change from Baseline (Week 1): Factor 2 Therapy-Related Problems | 2.78 (9.742) | -1.52 (15.841)
  IGSC: Epoch 2: Change from Baseline (Week 1): Factor 3 Therapy Setting | -6.48 (30.106) | 0.51 (11.773)
  IGSC: Epoch 2: Change from Baseline (Week 1): Factor 4 Treatment Costs | -9.72 (22.618) | 0.76 (31.282)
  IGSC: Epoch 3: Change from Baseline (Week 1): Factor 1 Treatment Interference: number analyzed (Participants) | 5 | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Factor 1 Treatment Interference | 4.17 (1.964) | 3.33 (4.120)
  IGSC: Epoch 3: Change from Baseline (Week 1): Factor 2 Therapy-Related Problems: number analyzed (Participants) | 5 | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Factor 2 Therapy-Related Problems | -14.58 (14.731) | 1.67 (14.613)
  IGSC: Epoch 3: Change from Baseline (Week 1): Factor 3 Therapy Setting: number analyzed (Participants) | 5 | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Factor 3 Therapy Setting | 19.44 (3.928) | 12.22 (16.387)
  IGSC: Epoch 3: Change from Baseline (Week 1): Factor 4 Treatment Costs: number analyzed (Participants) | 5 | 5
  IGSC: Epoch 3: Change from Baseline (Week 1): Factor 4 Treatment Costs | 0.00 (0.000) | 18.33 (40.139)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Factor 1 Treatment Interference | -2.78 (13.494) | -0.25 (13.046)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Factor 2 Therapy-Related Problems | -1.39 (9.001) | 1.14 (9.334)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Factor 3 Therapy Setting | 2.78 (16.005) | 4.55 (16.067)
  IGSC: Epoch 3: Change from Baseline (EOS/ET): Factor 4 Treatment Costs | 4.17 (16.672) | 14.39 (26.898)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (up to approximately 1.5 years)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Epoch 1: IGIV 200-600 mg/kg | Epoch 2: IGSC (20%) 50-200 mg/kg | Epoch 3: IGSC (20%) 100-400 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/7
Other Adverse Events (participants affected / at risk) | 11/17 | 16/17 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epoch 1: IGIV 200-600 mg/kg (N=17) | Epoch 2: IGSC (20%) 50-200 mg/kg (N=17) | Epoch 3: IGSC (20%) 100-400 mg/kg (N=7)
Myopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 3 | 1
Injection site erythema (General disorders) | 0 | 3 | 1
Injection site pain (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Vaccination site pain (General disorders) | 0 | 2 | 0
Administration site discolouration (General disorders) | 0 | 1 | 0
Administration site pain (General disorders) | 0 | 1 | 0
Administration site swelling (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Infusion site bruising (General disorders) | 0 | 1 | 0
Infusion site erythema (General disorders) | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 1 | 0
Infusion site pruritus (General disorders) | 0 | 1 | 0
Infusion site swelling (General disorders) | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Puncture site pain (General disorders) | 0 | 1 | 0
Vaccination site joint erythema (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic arthropathy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Occult blood positive (Investigations) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 3 | 1
Orthostatic intolerance (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT04346108/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT04346108/SAP_001.pdf